CLINICAL TRIAL: NCT05112081
Title: Evaluation of Botox Treatment in Patients With Chronic Scrotal Pain: a Randomized Double Blinded Control Trial
Brief Title: Evaluation of Botox Treatment on Chronical Scrotal Pain
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Nicolai Skov Schiellerup (Other)
Responsible Party: Sponsor-Investigator, Nicolai Skov Schiellerup, Principal investigator, Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-BTX-CSP
Record Dates: First submitted 2021-09-21; First posted 2021-11-08 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Scrotum Disease; Chronic Pain
Keywords: Chronical scrotal pain; CSP; Botox; BTX; minimal invasive procedure
MeSH Terms: conditions — Chronic Pain | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: This study is a prospective, randomized, placebo-controlled, double-blinded multi-center trial. Patients are included from the whole region of Southern Denmark.
  In case of successful spermatic cord block patients will be randomized to either BTX cord block or injection with sterile saline. Patients will be followed up according to the questionnaires. After three months, patients in the control arm will have the option to cross-over to the intervention arm.
Who Masked: Participant, Investigator
Masking Description: For randomization the research coordinator will place an information sheet containing the randomization in sealed envelopes (1:1 block randomization). At first treatment the research coordinator will open a sealed envelope revealing the randomization and prepare the solution needed. The patient and physician will be blinded for the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Botox injections (Experimental): Patients randomised to the intervention arm will be treated with injection of 100 units of botox in 10 ml sterile saline close to superficial inguinal ring.
  Interventions: Drug: Botulinum toxin type A
- Sterile saline injections (Placebo Comparator): Patients randomised to the control arm will be treated with injection of 10 ml sterile saline close to superficial inguinal ring.
  Interventions: Other: Sterile saline

INTERVENTIONS:
Drug: Botulinum toxin type A — The group will receive a solution of 100 units BTX with 10 ml sterile saline close to the superficial inguinal ring.
  Arms: Botox injections
Other: Sterile saline — The group will receive a solution of 10 ml sterile saline close to the superficial inguinal ring.
  Arms: Sterile saline injections

SUMMARY:
The aim of the study is to evaluate the effect of botox injections at the spermatic cord in patients with chronical scrotal pain.

A lot of patients experiences depressive symptoms and a lot feel isolated. The etiology if not fully understood and the condition poses a challenge for physicians.

The is no efficient minimal invasive treatment for these patients, and in severe cases patients are having there testicle removed.

By inject botox around the spermatic cord the investigators hope to relieve some of the pain in these patients and offer patients a new minimal invasive treatment.

The investigators aim to include 50 patients in this study, There will be randomised 1:1 to either the intervention arm (Botox) or control arm (sterile saline). Both patients and physicians will be blinded to the treatment.

Patients will undergo a thorough physical examination and will be asked to fill out questionaries to asses their quality of life.

After inclusion, patients will be followed closely for three months with physical examination and questionnaires.

After three months, patients in the control arm will have the opportunity to cross over to the intervention arm.

Data will be reported continuously.

DETAILED DESCRIPTION:
Background:

Chronic scrotal pain (CSP) is a common condition with a prevalence of 2.5-4.8% in male outpatients. Up to 40% of these patients report depressive symptoms and many feel isolated.

CSP is defined as intermittent or constant unilateral or bilateral scrotal pain with a significant impact on the patients daily life. The etiology of CSP is not fully understood but can be related to surgical procedures such as vasectomy, inguinal hernia repair, scrotal surgery and abdominal and groin surgery, even though no apparent cause can be identified in 25-50% of the cases.

When no obvious source of pain is found the most common approach usually begins with conservative treatment including analgesia, antibiotics and in some cases anticonvulsants and antidepressants. When conservative treatment fails, a minimal invasive procedure with local anesthesia cord block is often used before more invasive treatments such as denervation, vasovasostomy, orchiectomy or epididymectomy.

Of the minimally invasive procedures, spermatic cord block has proven to significantly reduce pain briefly in patients with CSP. Because of these findings, it has been proposed that a longer-lasting effect could be obtained with the use of OnabotulinumtoxinA (BTX). BTX is widely used in pain management in many painful diseases such as chronic pain syndrome, myofascial syndrome, headaches, arthritis, and neuropathic pain.

BTX interfere with neural transmission by blocking the release of acetylcholine, the principal neurotransmitter at the neuromuscular junction, causing muscle paralysis. Function can be recovered by the sprouting of nerve terminals and formation of new synaptic contacts which usually takes two to three months.

The use of BTX in patients with CSP have had varying results. One open-label study by Khambati et al reported a significant reduction in pain measured by VAS-score at follow-up after one and three months, but pain and tenderness had returned to baseline after six months. The only randomized double-blinded study by Dockray et al. showed no significant reduction in pain measured by VAS-score at follow-up after one month.

The aim of this study is to investigate the effect of chemical denervation with BTX injections on pain in patients with CSP.

Methods

Study population and recruitment Patients with CSP will be included according to the inclusion and exclusion criteria's (table 1). The following variables will be considered: gender, age, length of symptoms, and questionnaires, e.g., quality-of-life questionnaire (EQ-5D-5L) and Chronic Prostatitis Symptom Index (NIH-CPSI).

Determination of sample size Given that the true success rate for BTX, regarding the primary endpoint, is at least 0.70, and the placebo success rate among controls is 0.20. The investigators will need to study 23 experimental patients and 23 control patients to be able to reject the null hypothesis that the failure rates for experimental and control subjects are equal with probability (power) 0.9. The type I error probability associated with this test of this null hypothesis is 0.05. Considering potential dropouts, the investigators will include 25 patients per group.

Investigations Patients with CSP will undergo a comprehensive workup: including a thorough medical and psychical history, physical examination (i.e. inspection and palpation of penis, testis, funiculus, groin including inguinal channel, abdomen, direct rectal exploration with evaluation of the pelvic muscles, hips and column), investigations of lower urinary tract symptoms (i.e. uroflowmetry and bladder diary), blood work (i.e. creatinine, hematocrit, white blood cells count and C-reactive protein), Doppler ultrasonography of the scrotum, urine analyze (i.e. urine culture, test for chlamydia and gonorrhea). In case of no apparent cause, conservative treatment will be initiated with paracetamol 1000 mg four times a day, ibuprofen 400 mg three times a day or Prostazocin 2.5 mg three times a day. If no pain relief occurs within 30 days, patients are offered funicle cord block with 10 ml lidocaine 20 mg/ml. In case of a significant decrease in scrotal pain measured by VAS, patients will be offered inclusion in the study according to the study inclusion criteria and after written informed consent is provided.

Prior to BTX cord block patients will answer the following questionnaires:

1. Visual analog score for pain (VAS)
2. Quality-of-life (EQ-5D-5L)
3. Chronic Prostatitis Symptom Index (NIH-CPSI)
4. ICD-10 depression questionnaire (MDI)
5. Likert global assessment scale (L-GAS)
6. International Index of Erectile Function questionnaire (IIEF) Questionnaires will be repeated after 1, 2, 3, 4, 8 and 12 weeks. Physical examination will be repeated after 4, 8 and 12 weeks. Patients will be randomized to the intervention or control group.

In both groups injection of either BTX or sterile saline will be given close to the superficial inguinal ring. The intervention group will receive a solution of 100 IU BTX with 10 ml sterile saline while the control arm will receive 10 ml sterile saline. At the 3 months' time point, patients will be unblinded to the treatment and patients in the control group will have the option of cross-over.

Data analysis Univariate analysis and multivariate analysis will be performed: T-tests will be used to compare means between groups and chi-squared tests to compare dichotomous variables, and to adjust for unequal distribution of parameters at baseline, multivariate regression models, linear models in case of an interval scaled outcome, and logistic regression in case of a dichotomous outcome will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18 - 70 years
2. Unilateral or bilateral scrotal pain > 3 months
3. No other identifiable cause of pain
4. Insufficient effect of conservative treatment
5. A positive effect of local anesthesia spermatic cord block

Exclusion Criteria:

1. Inability to provide informed consent
2. Interest in trying to conceive with partner in the following 6 months
3. Local infection near the proposed injection site
4. History with an allergic reaction to BTX and / or human serum albumin
5. History of motor neuron disease or hemostatic disorder
6. Active urogenital cancer
7. Current use of botox injections which would result in a total dose of botox higher than 300 IE in the span of 3 months

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Effect on pain 3 months after treatment | 3 months
  Pain is evaluated on a Visual Analog Scale (VAS) from 0-10, where 0 is no pain and 10 is the maximal pain a patient can report.
  VAS prior to the treatment is compared to VAS 3 months after treatment.

SECONDARY OUTCOMES:
Duration of effect | 3 months
  Pain is evaluated on a Visual Analog Scale (VAS) from 0-10, where 0 is no pain and 10 is the maximal pain a patient can report.
  Patients will evaluate pain by VAS after 1, 2, 3, 4, 8 and 12 weeks
Changes in patient reported Quality of Life | 3 months
  Quality-of-life (EQ-5D-5L) Questionnaire containing 5 dimensions with a score scale from 0 - 5. A higher score correlates to a more negative impact on the patients life.
  Questionnaire will be repeated after 1, 2, 3, 4, 8 and 12 weeks
Changes in patient reported Quality of Life | 3 months
  Chronic Prostatitis Symptom Index (NIH-CPSI) The NIH-CPSI has a total score range from 0 to 43, and it includes three subscales addressing pain (score range 0-21).
  A higher score correlates to a more negative impact on the patients life.
  Questionnaire will be repeated after 1, 2, 3, 4, 8 and 12 weeks
Changes in patient reported Quality of Life | 3 months
  ICD-10 depression questionnaire (MDI) Patients can score 0 - 5 in multiple questions. A higher score signifies deeper depression.
  Questionnaire will be repeated after 1, 2, 3, 4, 8 and 12 weeks
Changes in patient reported Quality of Life | 3 months
  Likert global assessment scale (L-GAS) The scale is a rating scale for evaluating the overall functioning of the treatment. Patients can answer 0 - 100, where 100 is full satisfaction with the treatment.
  Questionnaire will be repeated after 1, 2, 3, 4, 8 and 12 weeks
Changes in patient reported Quality of Life | 3 months
  International Index of Erectile Function questionnaire (IIEF) Patients can score 0 - 5 and NA (not applicable). A lower score correlates to a more negative impact on the patients life.
  Questionnaire will be repeated after 1, 2, 3, 4, 8 and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mads H Poulsen, MD, PhD, Study Director — Assistant professor
Locations (1):
- Odense University Hospital, Odense C, Fyn, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data will be available at publication.
Supporting Information: Study Protocol
Time Frame: Will be available when patient enrolment starts and as long as the study is active.
Access Criteria: The protocol will be available to the public.

REFERENCES:
- [Background] Sigalos JT, Pastuszak AW. Chronic orchialgia: epidemiology, diagnosis and evaluation. Transl Androl Urol. 2017 May;6(Suppl 1):S37-S43. doi: 10.21037/tau.2017.05.23. PMID 28725616
- [Background] Schover LR. Psychological factors in men with genital pain. Cleve Clin J Med. 1990 Nov-Dec;57(8):697-700. doi: 10.3949/ccjm.57.8.697. PMID 2257677
- [Background] Aljumaily A, Forbes E, Al-Khazraji HAJ, Gordon A, Lau S, Jarvi KA. Frequency and severity of chronic scrotal pain in Canadian men presenting to urologists for infertility investigations. Transl Androl Urol. 2017 Dec;6(6):1150-1154. doi: 10.21037/tau.2017.11.28. PMID 29354503
- [Background] Singh V, Sinha RJ. Idiopathic chronic orchialgia - a frustrating issue for the clinician and the patient. Indian J Surg. 2008 Jun;70(3):107-10. doi: 10.1007/s12262-008-0032-x. Epub 2008 Jul 24. PMID 23133036
- [Background] Wu C, Jarvi K. Management of chronic scrotal content pain. Can Urol Assoc J. 2018 Jun;12(6 Suppl 3):S164-S166. doi: 10.5489/cuaj.5326. No abstract available. PMID 29875043
- [Background] Calixte N, Brahmbhatt J, Parekattil S. Genital pain: algorithm for management. Transl Androl Urol. 2017 Apr;6(2):252-257. doi: 10.21037/tau.2017.03.03. PMID 28540232
- [Background] Jarvi KA, Wu C, Nickel JC, Domes T, Grantmyre J, Zini A. Canadian Urological Association best practice report on chronic scrotal pain. Can Urol Assoc J. 2018 Jun;12(6):161-172. doi: 10.5489/cuaj.5238. Epub 2018 Feb 23. No abstract available. PMID 29485040
- [Background] Benson JS, Abern MR, Larsen S, Levine LA. Does a positive response to spermatic cord block predict response to microdenervation of the spermatic cord for chronic scrotal content pain? J Sex Med. 2013 Mar;10(3):876-82. doi: 10.1111/j.1743-6109.2012.02937.x. Epub 2012 Sep 27. PMID 23016953
- [Background] Kumar R. Therapeutic use of botulinum toxin in pain treatment. Neuronal Signal. 2018 Aug 31;2(3):NS20180058. doi: 10.1042/NS20180058. eCollection 2018 Sep. PMID 32714587
- [Background] Sim WS. Application of botulinum toxin in pain management. Korean J Pain. 2011 Mar;24(1):1-6. doi: 10.3344/kjp.2011.24.1.1. Epub 2011 Feb 25. PMID 21390172
- [Background] Colhado OC, Boeing M, Ortega LB. Botulinum toxin in pain treatment. Rev Bras Anestesiol. 2009 May-Jun;59(3):366-81. doi: 10.1590/s0034-70942009000300013. English, Portuguese. PMID 19488551
- [Background] Soares A, Andriolo RB, Atallah AN, da Silva EM. Botulinum toxin for myofascial pain syndromes in adults. Cochrane Database Syst Rev. 2014 Jul 25;2014(7):CD007533. doi: 10.1002/14651858.CD007533.pub3. PMID 25062018
- [Background] Moore C, Rackley R, Goldman H. Urologic applications of botox. Curr Urol Rep. 2005 Nov;6(6):419-23. doi: 10.1007/s11934-005-0035-0. PMID 16238914
- [Background] Aoki KR. Evidence for antinociceptive activity of botulinum toxin type A in pain management. Headache. 2003 Jul-Aug;43 Suppl 1:S9-15. doi: 10.1046/j.1526-4610.43.7s.3.x. PMID 12887389
- [Background] Nigam PK, Nigam A. Botulinum toxin. Indian J Dermatol. 2010;55(1):8-14. doi: 10.4103/0019-5154.60343. PMID 20418969
- [Background] Chancellor MB, Fowler CJ, Apostolidis A, de Groat WC, Smith CP, Somogyi GT, Aoki KR. Drug Insight: biological effects of botulinum toxin A in the lower urinary tract. Nat Clin Pract Urol. 2008 Jun;5(6):319-28. doi: 10.1038/ncpuro1124. Epub 2008 May 6. PMID 18461049
- [Background] Khambati A, Lau S, Gordon A, Jarvi KA. OnabotulinumtoxinA (Botox) nerve blocks provide durable pain relief for men with chronic scrotal pain: a pilot open-label trial. J Sex Med. 2014 Dec;11(12):3072-7. doi: 10.1111/jsm.12707. Epub 2014 Oct 6. PMID 25284738
- [Background] Dockray J, Aljumaily A, Lau S, Jarvi KA. A Randomized, Double-Blind, Controlled Trial Shows that Onabotulinum Toxin A Nerve Blocks do Not Provide Improved Pain Control in Men with Chronic Scrotal Pain. J Urol. 2020 Apr;203(4):767-772. doi: 10.1097/JU.0000000000000658. Epub 2019 Oct 18. PMID 31738115
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Heidenreich A, Olbert P, Engelmann UH. Management of chronic testalgia by microsurgical testicular denervation. Eur Urol. 2002 Apr;41(4):392-7. doi: 10.1016/s0302-2838(02)00023-4. PMID 12074809
- [Background] Park J, Park HJ. Botulinum Toxin for the Treatment of Neuropathic Pain. Toxins (Basel). 2017 Aug 24;9(9):260. doi: 10.3390/toxins9090260. PMID 28837075
- [Background] Lee CL, Kuo HC. Long-Term Efficacy and Safety of Repeated Intravescial OnabotulinumtoxinA Injections Plus Hydrodistention in the Treatment of Interstitial Cystitis/Bladder Pain Syndrome. Toxins (Basel). 2015 Oct 22;7(10):4283-93. doi: 10.3390/toxins7104283. PMID 26506388